## Signature Page for CR-AIR-008\_SAP Study CR-AIR-008 v2.0

| eSignature for Approval | Kun Wang |
|---|---|
| | Author 12-Dec-2018 09:48:40 GMT+0000 |
| eSignature for Approval | Annelies Legters |
| | Sponsor<br>12-Dec-2018 09:50:00 GMT+0000 |
| eSignature for Approval | Kees Meewisse |
| | Sponsor<br>12-Dec-2018 09:51:50 GMT+0000 |
| eSignature for Approval | Emmanuel Quinaux |
| | IDDI Statistician<br>13-Dec-2018 08:34:44 GMT+0000 |

Signature Page for CR-AIR-008\_SAP Study CR-AIR-008 v2.0



Version: 2.0

# **Statistical Analysis Plan**

| Sponsor: | Kiadis |
|---|---|
| Protocol Title: | An exploratory, open-label, multicenter study to evaluate the safety and efficacy of a two-dose regimen of ATIR101, a T-lymphocyte enriched leukocyte preparation depleted ex vivo of host alloreactive T-cells (using photodynamic treatment), in patients with a hematologic malignancy, who received a CD34-selected hematopoietic stem cell transplantation from a haploidentical donor |
| Study Code: | CR-AIR-008 |

| he undersigned certify that they have read, reviewed and approved this document. |
|---|
| Authors (IDDI): Katrien Verschueren, Senior Biostatistician Kun Wang, Senior Biostatistician |
| Approver (IDDI): Emmanuel Quinaux, Director Biostatistics |
| Sponsor Representative: Annelies Legters, Senior Director Clinical Operations |
| Signature and date |

TPL N°: eTPL SA-02-01 Of SOP SA-02.08 TPL Version: 02 

TPL Effective Date: 31 Mar 2016



## **Table of Contents**

| 1. L | IST OF ABBREVIATIONS AND DEFINITION OF TERMS | 4 |
|---|---|---|
| 2. I | NTRODUCTION | 6 |
| 3. 5 | STUDY DESIGN AND OBJECTIVES | 6 |
| | 3.1.1 Study Objective | 6<br>6<br>7 |
| 4. 6 | GENERAL ANALYSIS DEFINITIONS | 8 |
| 4.2<br>4.3<br>4<br>4<br>4 | A.1.1 Study Periods A.1.2 Visit Windows Planned analyses Definition of Populations A.3.1 Intention-To-Treat (ITT) Population A.3.2 Modified Intention-To-Treat (MITT) Population A.3.3 Per Protocol (PP) Population A.3.4 Safety Population Subgroup Definitions Calculated Variables Partial Dates Methods To Be Used For Handling Missing Data | 8 9 10 10 16 16 10 10 11 11 |
| 5. S | STUDY PATIENTS | 11 |
| 5.1<br>5.2<br>5.3 | Protocol Deviations | 12 |
| 6. E | DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS | 12 |
| 7. C | CONCOMITANT TREATMENT | 13 |
| 8. E | FFICACY EVALUATION | 13 |
| 8.1<br>8.2<br>8.3<br>8.4<br>8.5<br>8.6 | Secondary Endpoints Immune reconstitution Extent of Exposure Bone Marrow Biopsy / Aspirate | 13<br>14<br>14<br>15 |
| 9. S | SAFETY EVALUATION | 15 |
| 9.1<br>9.2<br>9.3<br>9.4<br>9.5 | Adverse Events Deaths and Serious Adverse Events Clinical Laboratory Determination | 16<br>17<br>17 |
| 10. | REFERENCES | 19 |

TPL Version: 02

### Kiadis - CR-AIR-008





#### Confidential

| 11. I | LIST OF TABLES/GRAPHS/LISTINGS | 23 |
|-------|--------------------------------|----|
| 11.1 | List of Statistical Tables | 23 |
| | List of Graphs | |
| 11 3 | List of Derived Data Listings | 27 |



## 1. List of Abbreviations and Definition of Terms

| Abbreviation | Term |
|--------------|---------------------------------------------------------------|
| AE | adverse event |
| ALT | alanine aminotransferase |
| AML | acute myeloid leukemia |
| ANC | absolute neutrophil count |
| AP | alkaline phosphatase |
| AST | aspartate aminotransferase |
| Ca | calcium |
| CD | cluster of differentiation |
| CI | chloride |
| CMV | cytomegalovirus |
| СТ | computed tomography |
| СТС | Common Terminology Criteria |
| DLT | dose-limiting toxicity |
| EBV | Epstein-Barr virus |
| ECG | electrocardiogram |
| ENT | ears, nose, throat |
| EU | European union |
| GCP | Good Clinical Practice |
| GRFS | GVHD-free, relapse-free survival |
| GVHD | graft-versus-host-disease |
| HBV | hepatitis B virus |
| HCT-CI | hematopoietic cell transplantation-specific comorbidity index |
| HCV | hepatitis C virus |
| HIV | human immunodeficiency virus |
| HLA | human leukocyte antigen |
| HSCT | hematopoietic stem cell transplantation |

Approved in Vault: 12/13/2018





| Abbreviation | Term |
|--------------|----------------------------------------------|
| HTLV | human T-lymphotropic virus |
| ICH | International Conference on Harmonization |
| ICF | informed consent form |
| Ig | immunoglobulin |
| ITT | intention-to-treat |
| LDH | lactate dehydrogenase |
| MCV | mean corpuscular volume |
| MedDRA | Medical Dictionary for Regulatory Activities |
| Mg | magnesium |
| MITT | modified intention-to-treat |
| MUGA | multiple gated acquisition |
| NCI | National Cancer Institute |
| NK | natural killer (cells) |
| os | overall survival |
| Р | phosphorus |
| PFS | progression-free survival |
| PP | per protocol |
| RBC | red blood cell |
| RRM | relapse-related mortality |
| SAE | serious adverse event |
| SAP | statistical analysis plan |
| TRM | transplant-related mortality |
| WBC | white blood cell |
| WHO | World Health Organization |
| WNV | West Nile virus |

TPL N°: eTPL SA-02-01 Of SOP SA-02.08 TPL Effective Date: 31 Mar 2016 TPL Version: 02 



Version: 2.0

#### 2. Introduction

This Statistical Analysis Plan was written for the clinical trial CR-AIR-008 conducted in EU and Canada. The ICH guideline E3 "Structure and Content of Clinical Study Reports" was used as a guide to the writing of the plan.

### 3. Study Design and Objectives

#### 3.1 Study Objectives

### 3.1.1 Study Objective

The study objective was to study the safety and efficacy of a repeat dose administration of ATIR101 in patients with a hematologic malignancy who received a T-cell depleted haploidentical hematopoietic stem cell transplantation (HSCT).

### 3.1.2 Study Endpoints

#### Primary safety endpoint

• The primary endpoint is the incidence of acute graft versus host disease (GVHD) grade III/IV up to 180 days post HSCT. Therefore, the primary analysis will be based on the data at 180 days after the HSCT.

#### Secondary endpoints (up to 12 months post HSCT)

- Incidence and severity of acute and chronic graft versus host disease (GVHD)
- Time to T-cell reconstitution, defined as the time to CD3+ in peripheral blood higher than  $0.2\times10^9/L$  (at two consecutive measurements; time to first measurement)
- Incidence and severity of viral, fungal, and bacterial infections
- Transplant-related mortality (TRM), defined as death due to causes other than disease relapse or progression, or other causes which are unrelated to the transplantation procedure (e.g. accident, suicide)
- Relapse-related mortality (RRM), defined as death due to disease relapse or disease progression
- Overall survival (OS), defined as the time from HSCT until death from any cause
- Progression-free survival (PFS), defined as the time from HSCT until relapse, disease progression, or death, whichever occurs first
- GVHD-free, relapse-free survival (GRFS), defined as the time from HSCT until acute GVHD grade III/IV, chronic GVHD requiring systemic treatment, relapse, or death, whichever occurs first



#### 3.2 Study Design

Study CR-AIR-008 is an exploratory, open-label, multicenter study. After signing informed consent, patients will receive an HSCT from a related, haploidentical donor, followed by a first ATIR101 infusion at a dose of  $2\times10^6$  viable T-cells/kg between 28 and 32 days after the HSCT. Patients will receive a second ATIR101 infusion at a dose of  $2\times10^6$  viable T-cells/kg between 70 and 74 days after the HSCT.

To evaluate safety of the second dose administration, the first 6 patients treated will be evaluated for the occurrence of dose-limiting toxicity (DLT), defined as acute GVHD grade III/IV within 120 days post HSCT (or within 42 days after the second ATIR101 infusion in case of prior dose delays). If within the first 6 patients no DLT is observed, treatment of the remaining 9 patients will continue with two ATIR101 doses of  $2\times10^6$  viable T-cells/kg. If within the first 6 patients at least 2 patients show DLT, the second ATIR101 infusion will be adjusted to a dose of  $1\times10^6$  viable T-cells/kg. If in one of the next 3 patients treated at this lower dose again DLT is observed, the second ATIR101 infusion will be halted and the remaining patients will be given only a single dose of ATIR101.

All patients treated with ATIR101 will be followed up until 12 months after the HSCT.

See **Appendix 1** for a detailed schedule of assessments.

### 3.3 Sample Size Justification

In total, 15 patients with a hematologic malignancy who are eligible for a haploidentical HSCT will be treated with two doses of ATIR101 (unless the second dose is halted for safety reasons). This sample size has been calculated with the following formula based on the primary endpoint (incidence of acute GVHD grade III/IV up to 180 days post HSCT):

$$n > \left(\frac{z^*}{m}\right)^2 p^* (1 - p^*)$$

Where:

n = sample size

 $z^*=z$ -value related to confidence interval, i.e. 1.645 for a one-sided 95% confidence interval

m = desired margin of error, i.e. 13%

 $p^* = \text{estimated population proportion, i.e. } 10\% \text{ acute GVHD grade III/IV } 180 \text{ days post HSCT}$ 

The primary endpoint is the incidence of acute GVHD grade III/IV up to 180 days post HSCT. Therefore, the primary analysis will be based on the data at 180 days after the HSCT. In the protocol it is defined that the study fails if the incidence of acute GVHD grade III/IV up to 180 days post HSCT in the MITT population exceeds 23%.

However, the above sample size calculation does not take into account that the number of patients meeting the primary endpoint is expected to be small (<10). Therefore, we cannot assume a normal distribution of proportions exists and exact statistics have to be applied.

For different data scenarios the upper limit of the one-side 70% confidence interval has been calculated with the Clopper-Pearson exact method using the R-package.

Approved in Vault: 12/13/2018



The y-value represents the number of "successes" (patients meeting the primary endpoint).

| conf. level<br>(power) | y (number of successes) | upper limit conf. interval (one-sided) |
|---|---|---|
| 70% | 0 | 0.077 |
| 70% | 1 | 0.155 |
| 70% | 2 | 0.228 |
| 70% | 3 | 0.299 |
| 70% | 4 | 0.368 |

The infusion of two doses of ATIR101 will be regarded safe for further clinical development if the upper limit of the one-sided confidence interval of the primary safety endpoint is below 23%. With a power of 70% and applying the Clopper-Pearson exact method, this corresponds to a maximum of 2 out of 15 patients in which acute GVHD grade III/IV within 180 days is observed. If the upper limit of the 70% confidence interval of the primary safety endpoint is above 23% (i.e. 3 or more out of 15 patients), the result of the study will be regarded indefinite and the study fails. In the latter case clinical development of the two-dose regimen will be halted.

### 4. General Analysis Definitions

Data will be analyzed using SAS (Version 9.3 or higher). Plots will be made in R.

As all patients will be treated with (one or two doses of) ATIR101, no tests of significance or no formal comparisons whatsoever will be carried out.

Descriptive statistics will be tabulated as follows:

- Categorical data will be summarized in contingency tables presenting frequencies and percentages.
- Continuous data will be summarized using number of non-missing values (n), mean, standard deviation, median, minimum and maximum values.

Moreover, the tables will be created by time point, as appropriate for the protocol or at a specified time point only if particularly specified. Listings are patient listings and ordered by patient id.

### 4.1 Study Period and Visit Window Definitions

### 4.1.1 Study Periods

ATIR101 was administered as one or two intravenous infusions. Patients treated with ATIR101 will be followed up until 12 months after the HSCT.

The end of the study is defined as the date at which the last data point from the last patient is received. In case it is decided that the study will be prematurely terminated, all patients who are still in the study should at least complete the visit at week 16 after the HSCT. After premature termination of the study, patients will be followed up for the occurrence of serious adverse events (SAEs) until 6 months after ATIR101 administration.

There are five distinct study periods:



- Screening period: period between informed consent & apheresis
- First treatment period: this period is divided in the following visits:
  - HSCT
  - Period between HSCT & ATIR101 infusion: weeks 1, 2 and 3
  - First ATIR101 infusion at week 4
- First follow-up period: weeks 5, 6, 7, 8 and 9
- Second treatment period: second ATIR101 infusion at week 10
- Second follow-up period: this period is divided in the following visits:
  - Weeks 11, 12, 13, 14, 15 and 16 (after HSCT)
  - Months 5, 6, 9 and 12 (after HSCT)

#### 4.1.2 Visit Windows

Visits must be performed within the following windows:

- Screening: between informed consent and apheresis
- HSCT (Day 0)
- Week 1: 1 week ± 2 days after the HSCT
- Week 2: 2 weeks ± 2 days after the HSCT
- Week 3: 3 weeks ± 2 days after the HSCT
- First ATIR101 infusion (Week 4): 28-32 days after the HSCT (unless postponed for medical reasons)
- Week 5: 5 weeks ± 2 days after the HSCT
- Week 6: 6 weeks ± 2 days after the HSCT
- Week 7: 7 weeks ± 2 days after the HSCT
- Week 8: 8 weeks ± 2 days after the HSCT
- Week 9: 9 weeks ± 2 days after the HSCT
- Second ATIR101 infusion (Week 10): 70-74 days after the HSCT but at least 42 days after the first ATIR101 infusion (unless postponed for medical reasons)
- Week 11: 11 weeks ± 2 days after the HSCT
- Week 12: 12 weeks ± 2 days after the HSCT
- Week 13: 13 weeks ± 2 days after the HSCT
- Week 14: 14 weeks ± 2 days after the HSCT
- Week 15: 15 weeks ± 2 days after the HSCT
- Week 16: 16 weeks ± 2 days after the HSCT
- Month 5: 5 months ± 1 week after the HSCT
- Month 6: 6 months ± 1 week after the HSCT
- Month 9: 9 months ± 2 weeks after the HSCT
- Month 12: 12 months ± 2 weeks after the HSCT



#### 4.2 Planned analyses

The final analysis will be performed when the last patient has been followed until 12 months after the HSCT or reached end of study.

### 4.3 Definition of Populations

All patients who provided informed consent and received an HSCT will be included in the analyses. The following analysis populations will be discerned:

#### 4.3.1 Intention-To-Treat (ITT) Population

The ITT population consists of all enrolled patients who received an HSCT whether or not they received ATIR101.

### 4.3.2 Modified Intention-To-Treat (MITT) Population

The MITT population consists of all ITT patients who received at least one dose of ATIR101. The primary analyses will be conducted using the MITT population.

### 4.3.3 Per Protocol (PP) Population

The PP population consists of all patients who:

- Received the first ATIR101 between 28 and 42 days after the HSCT,
- Received the second ATIR101 infusion between 70 and 84 days after the HSCT (if they received a second ATIR101 infusion),
- Showed hematologic engraftment (neutrophil count  $\geq 0.5 \times 10^9/L$  for 2 consecutive days and platelets  $\geq 20 \times 10^9/L$  for 3 consecutive days, without transfusion) at the time of the first ATIR101 infusion, and
- Did not present any major protocol deviations (see protocol Section 10.9).

All primary and secondary endpoint analyses will be remade using the PP population.

### 4.3.4 Safety Population

The Safety population will include all patients who received an HSCT and provided informed consent. Note that for this trial ITT and Safety populations are identical. ITT will be used for indicating population used (instead of Safety).

#### 4.4 Subgroup Definitions

Efficacy tables and graphs that will be made on ITT/ MITT/ PP population will be made for three groups: 1) all patients in the population 2) subgroup of patients that received one dose of ATIR101, and 3) subgroup of patients that received two doses of ATIR101. Safety tables that will be made on ITT / Safety population will be made for four groups: 1) patients that underwent HSCT and received single dose of ATIR101, 2) patients that underwent HSCT regardless of ATIR101, 3) subgroup of patients that received single dose of ATIR101, 4) subgroup of patients that received at least one dose of ATIR101. The different groups will be shown in the tables as different columns. Treatment Assignment and Treatment Arms are not applicable, as all patients will be treated with ATIR101.

#### 4.5 Calculated Variables

Study day 0 is defined as the day of HSCT procedure.



- The baseline for each variable is defined as the last assessment done in the screening period (between ICF and apheresis). Apheresis itself is part of baseline.
- Age is defined as follows: [(date of ICF)-(date of birth)+1]/365.25
- Event durations (e.g. AE duration) are calculated as follows: [end date start date +1]
- Time intervals (e.g. time from HSCT to ATIR101) are calculated as follows: [end date start date]
- Day of occurrence is calculated as follows: [event date -date of HSCT +1]

#### 4.6 Partial Dates

If part of the starting or ending dates of an adverse event (AE) is missing, the following convention will be used:

- For a missing day in an AE 'start date', the missing day is replaced by the first day of the month (e.g. UKMAY2003 -> 01MAY2003)
- For a missing day in an AE 'end date', the missing day is replaced by the last day of the month (e.g. UKMAR2003 -> 31MAR2003)

Missing AE intensities will not be imputed. Such AEs will be included in summaries by including a category of "missing" in the tables. If the assessment of the relationship of the AE to study medication is missing, we will assume that the AE is possibly related to study medication.

### 4.7 Methods To Be Used For Handling Missing Data

Any missing baseline values will not be imputed. If a subject has a missing baseline value that is required for a particular analysis, then the subject will be excluded from the statistical analysis.

Missing values will not be imputed for any time related endpoints. For patients who have not experienced the specific endpoints/events, the last known date of visit will be used as censoring time.

There will be no imputation of missing laboratory, vital sign, or ECG data.

#### 4.8 Changes to Protocol

This SAP is referring to amendment 1 of 20 November 2015 to original protocol from 9 July 2015.

### 5. Study Patients

#### **5.1** Disposition of Patients

The number of screened patients (who provided informed consent to the trial), the number of patients fulfilling in- and exclusion criteria, the number of enrolled patients (included in the study), the number of screen failures (including reason for screen failure), the number of patients who received an HSCT, the number of patients that discontinued before HSCT (including reason for discontinuation), the number of patients who received one dose of ATIR101, the number of patients who received two doses of ATIR101, the number of patients who discontinued after HSCT and before first ATIR101, after first ATIR101, and after second ATIR101 (including reason



for discontinuation) as well as the number of patients completing the study after first ATIR101 and after second ATIR101 will be summarized.

Individual patient disposition information will be listed additionally including details of 'other reason' if applicable, time from enrolment to apheresis, time from apheresis to HSCT, time from diagnosis (of first occurrence of hematologic malignancy) to HSCT, time from HSCT to ANC and Platelet engraftment, time from HSCT to first ATIR101 infusion, time from apheresis to first ATIR101 infusion and time from first till second ATIR101 infusion.

#### 5.2 Protocol Deviations

The major protocol deviations including an account of all identified major protocol deviations and other reasons for exclusion from the PP population (see 4.3.3. for definition of PP population) for the MITT population will be summarized. The details will be listed by patient. An additional listing will be made presenting all patients that are excluded from PP analysis (presenting patient ID, reason (protocol deviation or other), specification).

#### 5.3 In- and Exclusion Criteria

Listing of all in- and exclusion criteria not met will be provided.

### 6. Demographic and other Baseline Characteristics

Descriptive statistics with respect to patient and donor characteristics at baseline will be displayed for both the ITT and the MITT populations.

The variables to be summarized for patients are:

- Demographics: age, gender
- Hematologic malignancy and disease status: indications (AML, ALL, MDS), AML/ALL/MDS WHO classification level 1 and 2, FAB classification, disease status, number of previous remissions, EBMT risk score, Karnofsky score and HCT-CI ("Sorror score")

Patient cytogenetic abnormalities, molecular abnormalities, previous therapies as well as relevant medical history will be listed only.

The variables to be summarized for donors are:

- Demographics: age, gender, race and ethnicity; family relation between donor and patient
- HLA compatibility: mismatches at the HLA-A, -B and/or -DR loci (and if available at the HLA-C and -DQ loci) of the unshared haplotype will be assessed

An additional table with percentage of 3/6, 4/6, 5/6 and 6/6 matches based on HLA A, B and DR types for patients and donors and with percentage of x/8 and x/10 matches based on HLA A, B, C, DR and DQ types will be made. Assessment of matching (diploid, haploid) is made based on first two digits of both alleles per HLA type if only two digits are presented or if comparison is done between a two-digit result and a four-digit result. If the first two digits are equal, there is a match; otherwise a mismatch. If a four-digit result is compared to another four-digit result, all four digits must be identical in order to be a match. When one allele of an HLA type matches, it is called a haploid match. When two alleles match, it is called diploid match. These calculated x/6 and if available x/8 or x/10 scores will be added to the listing with patient and donor demographic information (i.e. age, gender, patient-donor relationship, HLA typing outcome and 2 scores).

TPL Effective Date: 31 Mar 2016



An additional listing depicting for patients the following information will be made: results of CT scan of the thorax (if applicable), echocardiogram or MUGA scan results (if applicable), results of pulmonary function test (if applicable), creatinine clearance results (if applicable), pregnancy test results (if applicable) and HIV-1, HIV-2, HBV, HCV, Treponema pallidum, HTLV-I (if tested), HTLV-II (if tested), WNV (if tested). In an additional listing the following donor data will be depicted: pregnancy test results (if applicable) and HIV-1, HIV-2, HBV, HCV, Treponema pallidum, HTLV-I (if tested), HTLV-II (if tested), WNV (if tested) results.

#### 7. Concomitant Treatment

All concomitant treatments will be summarized for the ITT population by WHO Drug code 2016, version 1 (using ATC classification) and listed.

### 8. Efficacy Evaluation

Efficacy evaluation will be performed on the MITT population. For the primary and secondary endpoints analyses (combination of efficacy and safety), sensitivity analyses will also be performed on the ITT and PP population.

#### 8.1 Primary Endpoint

The primary endpoint is the incidence of acute graft versus host disease (GVHD) grade III/IV up to 180 days post HSCT. Therefore, the primary analysis will be based on the data at 180 days after the HSCT. From the assumptions in Section 3.3 (Sample Size Justification) it can be derived that the study fails if the incidence of acute GVHD grade III/IV up to 180 days post HSCT in the MITT population exceeds 23% (desired margin of error + estimated population proportion). The proportion acute GVHD grade III/IV 180 days post HSCT will be calculated on all patients that received one or two doses ATIR101 combined only (as this is reflecting the sample size calculation).

#### 8.2 Secondary Endpoints

In this study the following secondary endpoints up to 12 months post HSCT have been identified:

- Incidence and severity of acute and chronic GVHD by time period. Time periods are defined as follows:
  - HSCT to first ATIR101 infusion
  - First ATIR101 infusion to 6 months post HSCT
  - 6 months to 1 year post HSCT
- Time from HSCT to T-cell reconstitution (i.e. the time to CD3+ in peripheral blood higher than 0.2x10<sup>9</sup>/L at two consecutive measurements; time to first measurement)
- Incidence and severity of viral, fungal, and bacterial infections by time period. Time periods are defined as follows:
  - Enrolment to HSCT
  - HSCT to first ATIR101 infusion
  - First ATIR101 infusion to 6 months post HSCT
  - 6 months to 1 year post HSCT



- Transplant-related mortality (TRM defined as death due to causes other than disease relapse or progression, or other causes which are unrelated to the transplantation procedure (e.g. suicide, accident)).
- Relapse-related mortality (RRM; defined as death due to disease relapse or disease progression).
- Overall survival (OS defined as the time from HSCT until death from any cause, or until last follow-up evaluation in the study for patients who were still alive.).
- Progression-free survival (PFS defined as the time from HSCT until relapse, disease progression, or death, whichever occurs first).
- GVHD-free, relapse free survival (GRFS), defined as the time until acute GVHD grade III/IV, chronic GVHD requiring systemic treatment, relapse, or death, whichever occurs first.

These endpoints will be analysed using descriptive statistics (tabulations for incidence and severity of viral, fungal and bacterial infections and GVHD). A separate summary for severe infections (grade 3/4/5) will also be made.

Time-related survival data (OS, PFS, GRFS) will be displayed with the Kaplan-Meier method. KM estimates at 6, and 12 months will also be provided. Time to event data will also be listed for the different survival endpoints (OS, PFS, GRFS). Times are displayed in months. Cumulative incidence curves taking into account competing risks will be used to display and estimate cumulative incidences of TRM (competing risk RRM), RRM (competing risk TRM), GVHD (competing risk death without GVHD) and time from HSCT to T-cell reconstitution (competing risk death without T-cell reconstitution).

If deemed necessary, comparison of the KM curves between the 1-dose group and the 2-dose group will be performed by using the log-rank test. The equality of cumulative incidence functions across patient groups will be tested using Gray's method (Gray 1988).

#### 8.3 Immune reconstitution

- Total lymphocytes and immunophenotyping on peripheral blood as measured by flow cytometry: CD3+ (T-cells), CD3+ CD8+ (cytotoxic T-cells), CD3+ CD4+ (helper T-cells), CD3- CD56+ (NK-cells), and CD19+ (B-cells)
- Immunoglobulins in peripheral blood: IgG, IgA, IgM

Total lymphocytes and immunophenotyping on peripheral blood as measured by flow cytometry: CD3+ (T-cells), CD3+ CD8+ (cytotoxic T-cells), CD3+ CD4+ (helper T-cells), CD3- CD56+ (NK-cells), and CD19+ (B-cells); and immunoglobulins in peripheral blood: IgG, IgA, IgM, will be summarized and listed. All CD measurements must be reported in absolute numbers of circulating lymphocytes (x10<sup>9</sup>/L). The listing is made as follows: by patient, parameters per category in columns and visits in rows. To the listing of immunoglobulins it will be added with \* if result is abnormal clinically not significant or with \*\* if abnormal clinically significant. For CD3+, CD3+ CD8+, CD3+ CD4+, CD3- CD56+, and CD19+, and for IgG, IgA and IgM a box plot with 25th and 75th percentiles (summarizing all data per available time point) will also be made.

#### 8.4 Extent of Exposure

Summary statistics will be made of the patient conditioning regimen (i.e. recommended TBI regimen, recommended non-TBI regimen, other) and HSCT



procedure: total amount of viable CD3+ cells/ $kg(x10^4)$  given to the patient and the total amount of viable CD34+ cells/ $kg(x10^6)$  given to the patient.

Four additional listings are made presenting for each patient: details on patient conditioning regimen, HSCT and first and second ATIR101 infusion. Variables presented but not limited to for patient conditioning regimen: conditioning regimen followed, medication name, start and stop date, dose and units and frequency. Variables presented for HSCT: date of HSCT, total amount of viable CD3+cells/kg(x10<sup>4</sup>) given to the patient and total amount of viable CD34+ cells/kg(x10<sup>6</sup>) given to the patient. Variables presented for first ATIR101 infusion: date of ATIR101 infusion with reason if not within 28-32 days after HSCT, number of days from HSCT, ATIR101 thawing interrupted Yes/No together with reason, start date/time of ATIR101 infusion, amount of ATIR101 infused, ATIR101 infusion interrupted Yes/No together with reason, etc. Variables presented for second ATIR101 infusion: date of ATIR101 infusion with reason if not within 70-74 days after HSCT, number of days from HSCT, ATIR101 thawing interrupted Yes/No together with reason, start date/time of ATIR101 infusion, amount of ATIR101 infused, ATIR101 infusion interrupted Yes/No together with reason, etc.

An additional table summarizing time from enrolment to apheresis, time from diagnosis to HSCT, time from apheresis to HSCT, time from HSCT to ANC and platelet engraftment, time from HSCT to first ATIR101 infusion, time from HSCT to second ATIR101 infusion, time from apheresis to first ATIR101 infusion and time from apheresis to second ATIR101 infusion will be made.

#### 8.5 Bone Marrow Biopsy / Aspirate

A table will summarize at the relevant time points (baseline, 6 months, 12 months and unscheduled visits) the amount and percentage of patients with myeloblasts <5% (Y/N) and the actual value of myeloblasts (in %) by bone marrow aspirate and biopsy separately.

A listing providing all details on bone marrow aspirate / biopsy will also be made.

#### 8.6 Engraftment and Chimerism

Engraftment is defined as neutrophil count  $\geq 0.5 \times 10^9/L$  for 2 consecutive days and platelets  $\geq 20 \times 10^9/L$  for 3 consecutive days. Time to ANC engraftment and platelet engraftment (from HSCT) will be summarized together with other time summaries (see 9.1). Chimerism results (i.e. total number of cells analysed, % donor cells, assessment done prior to ATIR101 infusion?) will be listed (including unscheduled visits).

#### 9. Safety Evaluation

The safety evaluation will be performed on the ITT population.

#### 9.1 DLT

To evaluate safety of the second dose administration, the first 6 patients treated will be evaluated for the occurrence of dose-limiting toxicity (DLT), defined as acute GVHD grade III/IV within 120 days post HSCT (or within 42 days after the second ATIR101 infusion in case of prior dose delays). If within the first 6 patients no DLT is observed, treatment of the remaining 9 patients will continue with two ATIR101 infusions of  $2\times10^6$  viable T-cells/kg. If within the first 6 patients at least 2 patients show DLT, the second ATIR101 infusion will be adjusted to a dose of  $1\times10^6$  viable T-cells/kg. If in one of the next 3 patients treated at this lower dose again DLT is observed, the second

TPL Effective Date: 31 Mar 2016



ATIR101 infusion will be halted and the remaining patients will be given only a single dose of ATIR101.

Details of the DLTs are presented in a listing.

#### 9.2 Adverse Events

Adverse events will be coded using MedDRA (Version 19.0).

For patients, adverse events (AEs) will be analyzed in terms of their type, incidence, severity and relationship to the study drug. An adverse event is treatment emergent if it is first observed or worsens on or after the date of first ATIR101 administration. In case of missing start date, the adverse event will be considered as treatment emergent. In listings it will be indicated if the AE is treatment emergent or not. If the event is ongoing at death, the event duration will be calculated using death date.

Tabulations of the number of patients who experienced AEs as well as severity of the events will be presented overall and by system organ class and preferred term. SOCs will be ordered by frequency (highest frequency first). PTs will be ordered alphabetically per SOC. Patients will only be counted once for each preferred term. In case a patient experienced the same event more than once, the worst severity will be presented. Both for AEs and SAEs, separate tables for ATIR101 related events only (defined as certainly, probably or possibly related or with missing relationship on AE form) will be made (by SOC and PT).

In addition, a summary table presenting an overview of all infection AEs from study entry (number/% of patients with at least one (S)AE, number/% of AEs with specific outcome, number/% of AEs per grade) will be provided. Number of events will also be indicated.

Tabulations of the number of donors who experienced (S)AEs as well as severity of the events will be presented overall and by system organ class and preferred term. Donors will only be counted once for each preferred term. In case a donor experienced the same event more than once, the worst severity will be presented.

A tabulation of AEs/SAEs will be made summarizing these events on the classification/category given (i.e. infection, relapse, GVHD, other etc.). Number of events will also be indicated.

For patients, the following AE listings will be made:

• GVHD AEs (including start since HSCT/ATIR101\*, outcome, duration, GVHD severity grade, NCI CTCAE severity grade, seriousness, causality).

The GVHD AE listing will contain the following detailed information: type, severity, organ involved (and score), number of days between start of GVHD and HSCT, number of days between start of GVHD and ATIR101\*, duration of GVHD in days, relation to ATIR101\*, action taken and outcome.

- Infection AEs (including type of infection, severity, seriousness, causality, details organism, start since HSCT/ATIR101\*, outcome, duration).
- Relapse AEs (including details on evaluation method, chimerism, start since HSCT/ATIR101\*, outcome, duration).
- Other AEs (including further information, severity, seriousness, causality, start since HSCT/ATIR101\*, outcome, duration).

<sup>\*</sup> Number of days between start of AE and first & second dose of ATIR101



• SAEs (type, reason for seriousness, duration, outcome)

For donors, a listing of all (S)AEs will be made.

#### 9.3 Deaths and Serious Adverse Events

Serious adverse events (SAEs) will be summarized by system organ class and preferred term.

Separate listings will detail all serious adverse events, graft failures / graft rejections and deaths, including number of days since HSCT/ATIR101\*, date and cause of death together with investigator classification of cause of death, during the study.

The number of deaths will be tabulated together with the primary cause of death. The details of the 'other cause' will be included in the listing.

### 9.4 Clinical Laboratory Determination

Hematology, blood chemistry and urinalysis parameters will be listed as follows: by patient, parameters per category in columns and visits in rows. Unscheduled visit results will be inserted based on the unscheduled visit's date. Results will be presented as e.g. 300 unit\*(L) or 850 unit\*\*(H). \*: abnormal not clinically significant; \*\*: abnormal clinically significant; L: if value below or equal to lower limit; H: if value above or equal to higher limit. For urinalysis only abnormal results are presented (result is abnormal based on the question (abnormal clinically (non-) significant?) or if outcome is not negative i.e. positive, traces, +, ++, etc.).

An additional listing presenting per patient and per parameter (hematology, blood chemistry, urinalysis) abnormal clinically significant values will also be made.

#### Table 1: List of safety laboratory tests

#### Hematology:

- Hematocrit
- Hemoglobin
- Mean corpuscular volume (MCV)
- Platelet count
- Red blood cell (RBC) count
- White blood cell (WBC) count
- Lymphocytes
- Monocytes
- Basophils
- Eosinophils
- Absolute neutrophil count (ANC)

#### <u>Urinalysis:</u>

• Bilirubin

#### **Blood Chemistry:**

- Albumin
- Alkaline phosphatase (AP)
- Alanine aminotransferase (ALT)
- Aspartate aminotransferase (AST)
- Calcium (Ca)
- Chloride (Cl)
- Creatinine
- Glucose
- Lactate dehydrogenase (LDH)
- Magnesium (Mg)
- Phosphorus (P)
- Potassium (K)
- Sodium (Na)
- Total bilirubin

Kiadis - CR-AIR-008 Version: 2.0



#### Confidential

| Glucose | Total protein |
|--------------------------------|---------------|
| • Ketones | • Urea |
| • Nitrite | |
| • Blood | |
| • pH | |
| • Protein | |
| • Specific gravity | |
| <ul> <li>Leukocytes</li> </ul> | |

### 9.5 CMV/EBV

CMV and EBV results are summarized in format of cross table (separate table for CMV and EBV). Overall (i.e. for all time points combined including unscheduled visits), for the donor/patient combinations with positive/positive, positive/negative, negative/positive and negative/negative baseline result, the percentage of patients with CMV/EBV outcome above the CMV/EBV limit at least one time point and below the CMV/EBV limit for all visits is presented.

In a listing, aVital Signs, Physical Findings and Other Observations Related to Safety Vital signs (respiration rate or oxygen saturation, temperature, weight, pulse rate, and supine blood pressure after 5 minutes of rest) will be listed.

Physical examination data (skin, ears/nose/throat (ENT), respiratory, cardiovascular, abdomen (including liver and spleen), and lymph nodes) will be listed.



### 10. References

Gray, R. (1988), "A Class of K-Sample Tests for Comparing the Cumulative Incidence of a Competing Risk," The Annals of Statistics, 16, 1141-1154.

SAS Statistical Analysis System. SAS Institute, Inc. Cary, NC, 1996.



### **Appendix 1: Schedule of Study Assessments**

| | Screening:<br>between<br>informed<br>consent &<br>apheresis | HSCT<br>(Day 0) | Week 1, 2, 3 | 1 <sup>st</sup> ATIR101 infusion Week 4 | Week 5, 6, 7, 8, 9 | 2 <sup>nd</sup> ATIR101 infusion Week 10 | Week<br>11, 12, 13,<br>14,15, 16 | Month 5, 6, 9, 12 |
|---|---|---|---|---|---|---|---|---|
| Informed consent patient and donor | X | | | | | | | |
| Apheresis patient and donor | X | | | | | | | |
| HSCT | | X | | | | | | |
| ATIR101 infusion | | | | X | | X | | |
| Patient characteristics and eligibility | | | | | | | | |
| Demographics | X | | | | | | | |
| Hematologic malignancy | X | | | | | | | |
| Medical history | X | | | | | | | |
| Performance status | X | | | | | | | |
| Physical examination | X | X | | X | X 1 | X | X <sup>2</sup> | |
| High resolution CT scan of the thorax | X <sup>3</sup> | | | | | | | |
| Echocardiogram/MUGA scan | X <sup>3</sup> | | | | | | | |
| Pulmonary function test | X <sup>3</sup> | | | | | | | |
| Creatinine clearance | X <sup>4</sup> | | | | | | | |
| Pregnancy test | X | | | | | | | |
| Viral testing | X | | | | | | | |

Only at Week 6 and Week 8

TPL N°: eTPL SA-02-01 TPL Version: 02 ****Of SOP SA-02.08

Only at Week 12, Week 14, and Week 16

If not already done within 6 weeks before signing informed consent

<sup>&</sup>lt;sup>4</sup> Calculated or measured, if not already done within 2 weeks before signing informed consent



| | Screening:<br>between<br>informed<br>consent &<br>apheresis | HSCT<br>(Day 0) | Week 1, 2, 3 | 1 <sup>st</sup><br>ATIR101<br>infusion<br>Week 4 | Week 5, 6, 7, 8, 9 | 2 <sup>nd</sup><br>ATIR101<br>infusion<br>Week 10 | Week<br>11, 12, 13,<br>14,15, 16 | Month 5, 6, 9, 12 |
|---|---|---|---|---|---|---|---|---|
| Donor characteristics and eligibility | | | T | <u> </u> | | | 1 | |
| Demographics | X | | | | | | | |
| HLA compatibility | X | | | | | | | |
| Pregnancy test | X | | | | | | | |
| Viral testing | X | | | | | | | |
| Donor adverse events | X | $\mathbf{X}^{1}$ | | | | | | |
| Vital signs | X | X | | X <sup>2</sup> | X | X <sup>2</sup> | X | |
| Safety laboratory tests | | | | | | | | |
| Hematology | X | X | X | X | X | X | X | |
| Blood chemistry | X | X | X | X | X | X | X | |
| Urinalysis | X | | | X | | X | X <sup>3</sup> | |
| CMV monitoring (PCR) | | X | X | X | X | X | X | X |
| EBV monitoring (PCR) <sup>4</sup> | | X | X | X | X | X | X | X |
| Engraftment | | | X | | | | | |
| Chimerism | | | | X 5 | | X 5 | | |

Until collection of stem cells

Before ATIR101 infusion. In addition, following ATIR101 infusion, pulse rate and supine blood pressure will be assessed after 15 minutes, 1, 2, 3, and 4 hours. Continuous oxygen monitoring will be done if the patient has respiratory problems.

Only at Week 16

If donor or patient is EBV positive before HSCT or as indicated Before ATIR101 infusion



| | Screening:<br>between<br>informed<br>consent &<br>apheresis | HSCT<br>(Day 0) | Week 1, 2, 3 | 1 <sup>st</sup> ATIR101 infusion Week 4 | Week 5, 6, 7, 8, 9 | 2 <sup>nd</sup> ATIR101 infusion Week 10 | Week<br>11, 12, 13,<br>14,15, 16 | Month 5, 6, 9, 12 |
|---|---|---|---|---|---|---|---|---|
| Efficacy and safety assessments | | | | | | | | |
| Immunophenotyping | X | | | X 1 | X <sup>2</sup> | X 1 | X | X |
| Immunoglobulins | X | | | X 1 | | X 1 | X <sup>3</sup> | X |
| Serum sampling <sup>4</sup> | X | X | | X 1 | X <sup>2</sup> | X 1 | X | X |
| Peripheral blood sampling <sup>5</sup> | | | | | X 6 | | X 6 | X 6 |
| Infection assessment | X | X | X | X | X | X | X | X |
| Disease assessment <sup>7</sup> | X | X | X | X | X | X | X | X |
| GvHD assessment | | | X | X | X | X | X | X |
| Mortality | | Continuous recording | | | | | | |
| Other adverse events | X | X | X | X | X | X | X | |
| Serious adverse events | | Continuous recording | | | | | | |
| Concomitant medications | X | X | X | X | X | X | X | X |

- Before ATIR101 infusion
- Only at Week 5, Week 7, and Week 9
- Only at Week 11, Week 13, and Week 16
- For measuring cytokine levels and/or immunoglobulins against specific antigens
- For measuring pathogen-specific T-cells
- Only at Week 6, Week 12, Month 6, and Month 12
- Includes bone marrow aspirate and/or biopsy at Screening, Month 6 and 12 after HSCT unless relapse has already been confirmed, and in case of suspected relapse



## 11. List of Tables/Graphs/Listings

### 11.1 List of Statistical Tables

| Number | Description | Population |
|---|---|---|
| Table 14.01.01 | Patient disposition | All patients |
| Table 14.01.02 | Summary of major protocol deviations and other reasons for exclusion from the PP population | MITT |
| Table 14.01.03 | Patient demographics | ITT, MITT |
| Table 14.01.04 | Patient baseline disease characteristics | ITT, MITT |
| Table 14.01.05 | Donor demographics | ITT, MITT |
| Table 14.01.06 | Matching score based on HLA typing patient - donor | ITT, MITT |
| Table 14.01.07 | Concomitant medications | ITT |
| Table 14.01.08 | Summary of durations | ITT, MITT |
| Table 14.02.01 | Incidence of acute graft versus host disease (GVHD) grade III/IV up to 180 days post HSCT | MITT, ITT, PP |
| Table 14.02.02.01 | Incidence and severity of acute and chronic GVHD by time period | MITT, ITT, PP |
| Table 14.02.02.02 | Incidence and severity of viral, fungal, and bacterial infections by time period | MITT, ITT, PP |
| Table 14.02.02.03 | KM estimates of OS (at 6 and 12 months) | MITT, ITT, PP |
| Table 14.02.02.04 | KM estimates of PFS (at 6 and 12 months) | MITT, ITT, PP |
| Table 14.02.02.05 | KM estimates of GRFS (at 6 and 12 months) | MITT, ITT, PP |
| Table 14.02.03.01 | Cumulative incidence of TRM (cumulative incidence function) | MITT, ITT, PP |
| Table 14.02.03.02 | Cumulative incidence of RRM (cumulative incidence function) | MITT, ITT, PP |
| Table 14.02.03.03 | Cumulative incidence of GVHD (cumulative incidence function) | MITT, ITT, PP |

Approved in Vault: 12/13/2018



Version: 2.0

| Table 14.02.03.04 | Cumulative incidence of T-cell reconstitution (cumulative incidence function) | MITT, ITT, PP |
|---|---|---|
| Table 14.02.04 | Immune reconstitution (immunophenotyping and immunoglobulins) | MITT, |
| Table 14.02.05 | Extent of exposure | MITT |
| Table 14.02.06 | Engraftment and Chimerism | MITT |
| Table 14.02.07 | Bone marrow aspirate | MITT |
| Table 14.03.01.01 | Patient adverse events summary | ITT |
| Table 14.03.01.02 | Patient adverse events by SOC and PT | ITT |
| Table 14.03.01.03 | Patient adverse events by SOC, PT and severity | ITT |
| Table 14.03.01.04 | Patient ATIR101 related adverse events by SOC and PT | ITT |
| Table 14.03.01.05 | Patient treatment-emergent adverse events by SOC and PT | ITT |
| Table 14.03.01.06 | Patient treatment-emergent adverse events by SOC, PT and severity | ITT |
| Table 14.03.02.01 | Patient serious adverse events summary | ITT |
| Table 14.03.02.02 | Patient serious adverse events by SOC and PT | ITT |
| Table 14.03.02.03 | Patient serious adverse events by SOC, PT and severity | ITT |
| Table 14.03.02.04 | Patient ATIR101 related serious adverse events by SOC and PT | ITT |
| Table 14.03.02.05 | Patient treatment-emergent serious adverse events by SOC and PT | ITT |
| Table 14.03.02.06 | Patient treatment-emergent serious adverse events by SOC, PT and severity | ITT |
| Table 14.03.03 | Overview of all patient infection adverse events | ITT |
| Table 14.03.04.01 | Donor adverse events by SOC and PT | ITT |
| Table 14.03.04.02 | Donor adverse events by SOC, PT and severity | ITT |
| Table 14.03.05 | Deaths | ITT |
| Table 14.03.06 | CMV/EBV summary | ITT |





Note: if a table needs to be made on several populations e.g. MITT and ITT the table numbering is as follows: Table 14.x.x.1 and Table 14.x.x.2.



## 11.2 List of Graphs

| Number | Description | Population |
|--------------------|------------------------------------|---------------|
| Figure 14.02.01 | Kaplan-Meier plot PFS | MITT, ITT, PP |
| Figure 14.02.02 | Kaplan-Meier plot OS | MITT, ITT, PP |
| Figure 14.02.03 | Kaplan-Meier plot GRFS | MITT, ITT, PP |
| Figure 14.02.04 | Cumulative incidence curve of TRM | MITT, ITT, PP |
| Figure 14.02.05 | Cumulative incidence curve of RRM | MITT, ITT, PP |
| Figure 14.02.06 | Cumulative incidence curve of GVHD | MITT, ITT, PP |
| Figure 14.02.07.01 | Box-plot for lymphocytes | MITT |
| Figure 14.02.07.02 | Box-plot for CD3+ | MITT |
| Figure 14.02.07.03 | Box-plot for CD3+ CD8+ | MITT |
| Figure 14.02.07.04 | Box-plot for CD3+ CD4+ | MITT |
| Figure 14.02.07.05 | Box-plot for CD3- CD56+ | MITT |
| Figure 14.02.07.06 | Box-plot for CD19+ | MITT |
| Figure 14.02.07.07 | Box-plot for IgG | MITT |
| Figure 14.02.07.08 | Box-plot for IgM | MITT |
| Figure 14.02.07.09 | Box-plot for IgA | MITT |

Note: if a figure needs to be made on several populations e.g. MITT and ITT/PP, the figure numbering is as follows: Figure 14.x.x.1 and Figure 14.x.x.2.

Approved in Vault: 12/13/2018



### 11.3 List of Derived Data Listings

Notes: Listings will be produced on ALL patients, and sorted by patient ID. The patient ID will be followed by one of the letters below (i.e. a, b, c, d, or e) to indicate if patient belongs to:

- (a) MITT single dose
- (b) MITT double dose
- (c) ITT single dose (no MITT)
- (d) Screening failure
- (e) No HSCT (no screening failure)

And this list will be put in a footnote.

| Number | Description | Population |
|---|---|---|
| Listing 16.02.01 | Patient disposition | All patients |
| Listing 16.02.02 | Durations (including time to engraftment) | All patients |
| Listing 16.02.03 | Major protocol deviations | All patients |
| Listing 16.02.04 | Patients excluded from per-protocol population | All patients |
| Listing 16.02.05 | In- and exclusion criteria not met | All patients |
| Listing 16.02.06 | Patient and donor demographics | All patients |
| Listing 16.02.07 | Patient and donor baseline CMV/EBV | All patients |
| Listing 16.02.08 | Patient baseline disease characteristics | All patients |
| Listing 16.02.09 | Additional patients baseline disease characteristics (CT, ECG, pulmonary, creatinine, pregnancy, virology) | All patients |
| Listing 16.02.10 | Patient cytogenetic abnormalities | All patients |
| Listing 16.02.11 | Patient molecular abnormalities | All patients |
| Listing 16.02.12 | Patient previous therapies | All patients |

Approved in Vault: 12/13/2018

TPL N°: eTPL SA-02-01 TPL Version: 02 ****Of SOP SA-02.08



| Listing 16.02.13 | Patient medical history | All patients |
|---|---|---|
| Listing 16.02.14 | Concomitant medications | All patients |
| Listing 16.02.15 | PFS: time to event data | All patients |
| Listing 16.02.16 | OS: time to event data | All patients |
| Listing 16.02.17 | GRFS: time to event data | All patients |
| Listing 16.02.18 | Details of patient conditioning regimen | All patients |
| Listing 16.02.19 | Details of HSCT procedure | All patients |
| Listing 16.02.20 | Details of ATIR101 infusion | All patients |
| Listing 16.02.21 | Bone marrow aspirate | All patients |
| Listing 16.02.22 | Engraftment and Chimerism | All patients |
| Listing 16.02.23 | DLTs | All patients |
| Listing 16.02.24 | GVHD adverse events (patients) | All patients |
| Listing 16.02.25 | Infection adverse events (patients) | All patients |
| Listing 16.02.26 | Relapse adverse events (patients) | All patients |
| Listing 16.02.27 | Other adverse events (patients) | All patients |
| Listing 16.02.28 | Serious adverse events (patients) | All patients |
| Listing 16.02.29 | All adverse events (donors) | All patients |
| Listing 16.02.30 | Deaths (including graft failures / graft rejections) | All patients |
| Listing 16.02.31 | Graft failures / graft rejections | All patients |
| Listing 16.02.32 | Immune reconstitution (immunophenotyping and immunoglobulins) | All patients |
| Listing 16.02.33 | Laboratory data for hematology | All patients |
| Listing 16.02.34 | Laboratory data for serum chemistry | All patients |



Version: 2.0

| Listing 16.02.35 | Urinalysis data | All patients |
|---|---|---|
| Listing 16.02.36 | Per patient listing with clinically significant abnormal lab values (hematology, blood chemistry, urinalysis) | All patients |
| Listing 16.02.37 | Patient CMV/EBV | All patients |
| Listing 16.02.38 | Vital signs | All patients |
| Listing 16.02.39 | Physical examinations | All patients |